CLINICAL TRIAL: NCT04562402
Title: Phacoemulsification With Endoscopic Cyclophotocoagulation vs Phacoemulsification Alone in Primary Angle Closure (PHEPHA): A Randomized Clinical Trial
Brief Title: Phaco-ECP vs Phaco Alone in Primary Angle Closure
Acronym: PHEPHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Principal Investigator, Adi Al Owaifeer, MBBS, Consultant, King Khaled Eye Specialist Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1956-P
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Glaucoma, Angle-Closure
Keywords: Glaucoma; Endoscopic cyclophotocoagulation; Laser; Intraocular pressure; Phacoemulsification; Primary angle closure glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure; Glaucoma | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phacoemulsification with endoscopic cyclophotocoagulation (Active Comparator): Cataract extraction via phacoemulsification along with endoscopic cyclophotocoagulation of the ciliary body.
  Interventions: Procedure: Phacoemulsification; Procedure: Endoscopic cyclophotocoagulation
- Phacoemulsification alone (Active Comparator): Cataract extraction via phacoemulsification.
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — cataract surgery via phacoemulsification
Procedure: Endoscopic cyclophotocoagulation — Endoscopic ablation of the ciliary body
  Arms: Phacoemulsification with endoscopic cyclophotocoagulation

SUMMARY:
Comparison between phacoemulsification with endoscopic cyclophotocoagulation versus phacoemulsification alone in patients with either primary angle closure or primary angle closure glaucoma presenting with cataract or a clear lens.

DETAILED DESCRIPTION:
The purpose of our current randomized clinical trial is to compare phacoemulsification with endoscopic cyclophotocoagulation (PHE) versus phacoemulsification alone (PHA) in patients with either primary angle closure (PAC) or primary angle closure glaucoma (PACG) presenting with cataract or a clear lens.

ELIGIBILITY:
Inclusion Criteria:

1. Age is above 40 years old.
2. A diagnosis of either PAC or PACG. PAC will be defined as the presence of irido-trabecular contact on gonioscopy, either appositional or in the presence of peripheral anterior synechiae (PAS), without indentation (or prior documentation before a LPI has been performed) without any evidence of glaucomatous optic neuropathy. PACG will be defined as PAC along with an evidence of glaucomatous optic neuropathy. An optic neuropathy secondary to glaucoma will be defined as evidence of structural and functional damage suggestive of glaucoma as demonstrated by clinical examination, optical coherence tomography, and visual field testing.
3. IOP measurement that is more than 21 mmHg (not exceeding 35 mmHg) without the use of glaucoma medications or less than 21 mmHg with medications.
4. Patient is able to give an informed consent and tolerate a period of medication washout.

Exclusion Criteria:

1. Previous intraocular surgery (including CPC). Glaucoma laser procedures are allowed (e.g. LPI, iridoplasty, and laser trabeculoplasty).
2. Previous ocular trauma.
3. A central corneal thickness that does not lie between 500 and 600 microns.
4. A diagnosis of nanophthalmos (defined as an axial length that is less than 20 mm).
5. Presence of pseudoexfoliation.
6. Presence of secondary causes of angle closure such as neovascular glaucoma and uveitic glaucoma.
7. Presence of diabetic retinopathy (active PDR or active DME) or agerelated macular degeneration. PHEPHA Protocol Version 2 September 3, 2020
8. Advanced glaucoma as defined by the Glaucoma Severity Staging System12 (mean deviation worse than -12.01 dB and at least one of the following: 1. On pattern deviation plot, greater than or equal to 50% but fewer than 75% of points depressed below the 5% level and greater than or equal to 25% but fewer than 50% of points depressed below 1% level 2. Any point within central 5 degrees with sensitivity < 0db 3. Both hemifields containing a point(s) with sensitivity < 15 dB within 5 degrees of fixation).
9. Any ocular or systemic condition that is presumed to prevent reliable clinical examination and/or visual field testing.
10. Pregnancy.
11. Inability to attend postoperative follow ups for a period of 12 months after surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-08-16 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | 12 months
  Change in IOP between baseline (pre-intervention) and the last follow-up visit
Number of glaucoma medications | 12 months
  Change in the number of glaucoma medications between baseline (pre-intervention) and the last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Adi Al Owaifeer, MBBS, Principal Investigator — King Khaled Eye Specialist Hospital; Ibrahim Alobaida, MD, Principal Investigator — King Khaled Eye Specialist Hospital
Locations (1):
- King Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided